CLINICAL TRIAL: NCT07359950
Title: Effects of Film-Based Music Therapy With LLM-Generated Culturally Adapted Verbal Suggestions on Anxiety, Affect, and Heart Rate Among Chinese Young Adults: A Randomized Controlled Trial
Brief Title: Film-Based Music Therapy With AI-Generated Verbal Guidance for Anxiety in Young Adults
Acronym: EAST-MUSIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wen Li (Other)
Responsible Party: Sponsor-Investigator, Wen Li, Principal Investigator, Universiti Sains Malaysia
Organization: Universiti Sains Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: USM-JEPeM-22120811; USM/JEPeM/22120811 (Registry Identifier: Universiti Sains Malaysia Human Research Ethics Committee (JEPeM))
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Anxiety; Psychological Stress; Emotional Regulation
Keywords: Music therapy; Verbal suggestions; Artificial intelligence; Large language models; Cultural adaptation; Eastern aesthetic imagery; University students; Heart rate variability
MeSH Terms: conditions — Anxiety Disorders; Stress, Psychological; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of three parallel groups and receive a single music-based intervention according to group assignment.
Masking Description: This study is conducted as an open-label trial. Due to the nature of the music-based interventions and verbal guidance, neither participants nor investigators are blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Eastern Imagery Music Therapy Group (Experimental): Participants assigned to this arm listen to a curated music program accompanied by verbal guidance generated by a large language model. The verbal guidance is designed to evoke Eastern aesthetic imagery and is delivered during a single 25-30 minute music listening session.
  Interventions: Behavioral: Music Listening With AI-Generated Eastern Imagery Verbal Guidance
- Standard Music Therapy Group (Active Comparator): Participants assigned to this arm listen to music accompanied by standard relaxation-oriented verbal guidance commonly used in music therapy practice. The intervention is delivered during a single 25-30 minute music listening session.
  Interventions: Behavioral: Music Listening With Standard Verbal Guidance
- Music-Only Relaxation Group (Active Comparator): Participants assigned to this arm listen to relaxing music without any verbal guidance during a single 25-30 minute session.
  Interventions: Behavioral: Music-Only Relaxation

INTERVENTIONS:
Behavioral: Music Listening With AI-Generated Eastern Imagery Verbal Guidance — Participants listen to a curated music program accompanied by verbal guidance generated by a large language model. The verbal guidance is designed to evoke Eastern aesthetic imagery and is delivered by a researcher during a single 25-30 minute music listening session in a quiet setting.
  Arms: Eastern Imagery Music Therapy Group
Behavioral: Music Listening With Standard Verbal Guidance — Participants listen to music accompanied by standard relaxation-oriented verbal guidance commonly used in music therapy practice. The guidance is delivered during a single 25-30 minute music listening session in a quiet setting.
  Arms: Standard Music Therapy Group
Behavioral: Music-Only Relaxation — Participants listen to relaxing music without any verbal guidance during a single 25-30 minute session in a quiet setting.
  Arms: Music-Only Relaxation Group

SUMMARY:
This study aims to examine whether music-based relaxation combined with different types of verbal guidance can help reduce anxiety and improve emotional well-being in young adults.

University students often experience high levels of stress related to academic demands and daily life. Music listening is commonly used as a simple and safe method to promote relaxation. In addition to music itself, verbal guidance during music listening may influence how individuals imagine, interpret, and emotionally respond to the music experience.

In this study, participants are randomly assigned to one of three groups. One group listens to music accompanied by verbal guidance generated by a large language model and designed to reflect Eastern aesthetic imagery. A second group listens to music with standard relaxation guidance commonly used in music therapy. A third group listens to relaxing music without any verbal guidance. Each participant takes part in a single music listening session lasting approximately 25-30 minutes.

Levels of anxiety, positive and negative emotions, and heart rate are measured before and after the music session. By comparing the results across the three groups, this study seeks to better understand whether culturally adapted verbal guidance can enhance the effects of music-based relaxation for young adults.

DETAILED DESCRIPTION:
This study is a single-center, randomized controlled trial designed to investigate the effects of music-based interventions with different types of verbal guidance on anxiety and emotional regulation in young adults.

Eligible university students are recruited and randomly assigned in equal numbers to one of three parallel groups: (1) a music intervention with verbal guidance generated by a large language model and designed to evoke Eastern aesthetic imagery; (2) a standard music therapy condition that includes conventional relaxation-oriented verbal suggestions; and (3) a music-only relaxation condition without verbal guidance. Randomization is conducted using a simple random allocation procedure.

All participants complete baseline assessments prior to the intervention. Each participant then takes part in a single music listening session lasting approximately 25-30 minutes in a quiet classroom setting. During the session, participants are seated comfortably with eyes closed and instructed to listen attentively to the music. Verbal guidance, when present, is delivered by a researcher during the music session.

Primary and secondary outcomes are assessed immediately before and after the intervention. Anxiety is measured using a standardized self-report anxiety scale. Emotional states are assessed using validated measures of positive and negative affect. Heart rate is recorded as an objective physiological indicator of autonomic arousal using a smartphone-based photoplethysmography method.

This study aims to provide empirical evidence on whether culturally adapted verbal guidance, generated by artificial intelligence, can enhance the psychological and physiological effects of music-based relaxation in young adults.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 25 years at the time of enrollment.
* Currently enrolled as a university student.
* Able to understand the study procedures and provide written informed consent.
* Willing to participate in a single music listening session lasting approximately 25-30 minutes.
* Able to complete self-report questionnaires before and after the intervention.

Exclusion Criteria:

* Self-reported history of diagnosed psychiatric disorders (e.g., major depressive disorder, anxiety disorders, psychotic disorders).
* Current use of psychotropic medications that may significantly affect mood or anxiety.
* Self-reported hearing impairment that could interfere with music listening.
* Self-reported cardiovascular conditions or other medical conditions that could affect heart rate measurements.
* Participation in other psychological or behavioral intervention studies within the past 30 days.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 123 (Actual)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-01-30 (Actual); Study Completion 2026-01-30 (Actual)

PRIMARY OUTCOMES:
Change in State Anxiety Score | Immediately before and immediately after the single 25-30 minute music listening session
  State anxiety is assessed using the State subscale of the State-Trait Anxiety Inventory (STAI-S), a validated self-report questionnaire consisting of 20 items. Scores range from 20 to 80, with higher scores indicating greater state anxiety. The primary outcome is the change in STAI-S score from before to immediately after the intervention.

SECONDARY OUTCOMES:
Change in Positive Affect Score | Immediately before and immediately after the single 25-30 minute music listening session
  Positive affect is measured using the Positive Affect subscale of the Positive and Negative Affect Schedule (PANAS). The subscale consists of 10 items assessing positive emotional states, with higher scores indicating greater positive affect. The outcome is defined as the change in positive affect score from before to immediately after the intervention.
Change in Negative Affect Score | Immediately before and immediately after the single 25-30 minute music listening session
  Negative affect is measured using the Negative Affect subscale of the Positive and Negative Affect Schedule (PANAS). The subscale consists of 10 items assessing negative emotional states, with higher scores indicating greater negative affect. The outcome is defined as the change in negative affect score from before to immediately after the intervention.
Change in Heart Rate | Immediately before and immediately after the single 25-30 minute music listening session
  Heart rate is recorded as an objective physiological indicator of autonomic arousal using a smartphone-based photoplethysmography method. The outcome is defined as the change in mean heart rate measured immediately before and immediately after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Wen Li, PhD, Principal Investigator — Aba Teachers College
Locations (1):
- Aba Teachers College, Aba, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided